CLINICAL TRIAL: NCT06832657
Title: A Randomized, Double-blind, Placebo-controlled Phase 1 Study of JMKX003948 Ophthalmic Suspension to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Dose(s) in Healthy Participants
Brief Title: Study of JMKX003948 Ophthalmic Suspension in Healthy Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JMKX003948-101
Record Dates: First submitted 2024-12-25; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Age-Related Macular Degeneration (AMD); Diabetic Macular Edema (DME)
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JMKX003948 Ophthalmic Suspension (Experimental)
  Interventions: Drug: JMKX003948 Ophthalmic Suspension
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JMKX003948 Ophthalmic Suspension — JMKX003948 Ophthalmic Suspension with formulation 1% (15 mg/1.5 mL), 2% (30 mg/1.5 mL), 3% (45 mg/1.5 mL), 5% (75 mg/1.5 mL)
  Arms: JMKX003948 Ophthalmic Suspension
Drug: Placebo — JMKX003948 Ophthalmic Suspension placebo
  Arms: Placebo

SUMMARY:
The study is a randomized, double-blind, placebo-controlled, phase 1 study of JMKX003948 Ophthalmic Suspension to evaluate the safety, tolerability and PK of single and multiple ascending doses in healthy participants.

Participant will be randomized to receive either JMKX003948 Ophthalmic Suspension (1%, 2%, 3% or 5%) or matching placebo (JMKX003948 Ophthalmic Suspension: placebo= 6: 2, N=8 per cohort).

Five cohorts (Cohort 1-5) are planned. Cohorts could also de-escalate to a lower concentration if current formulation was not tolerated (Cohort 1b, 2b and 3b). In case of de-escalation, Cohort 1b and 2b will continue to escalate to Cohort 1c and Cohort 2c, respectively.

Participants will be admitted to the site on Day -1 after screening (up to 28 days), and remain domiciled until Day 14 for Cohort 1-4, Day 8 for other cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males and/or females, 18 to 45 years of age (inclusive) at the date of signed consent form.
2. Body mass index (BMI) greater than or equal to 18 and less than 32 (kg/m2) and a minimum body weight of 45 kg.
3. Able to participate and comply with all study procedures and restrictions, and willing to provide written informed consent to participate in the study.
4. Women of child-bearing potential and sexually active males willing to use highly effective methods of contraception from screening until 3 months after last dose of study drug. In addition, participants must not donate sperm/egg for the time period specified above.

Exclusion Criteria:

1. History of disease of ocular surface, fundus, central nervous system, psychiatric and psychological condition, cardiovascular system, kidney, liver, digestive system, respiratory system, or metabolic/endocrine system, or other disease that in the opinion of the Investigator (or medically qualified designee) may make participation unsafe for the participant or interfere with study evaluations.
2. Any abnormal examination with clinical significance may interfere with study evaluations in opinion of the Investigator (or medically qualified designee).
3. History of eye trauma or surgery including LASIK/LASEK.
4. Any corrected visual acuity < 20/20, or intraocular pressure ≥ 21 mmHg.
5. Clinically significant abnormalities on ophthalmic examination that would hinder the assessment of the eye or data collection at the discretion of the Investigator and/or ophthalmologist (or medically qualified designee).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | From Day1 to up to Day14
  Incidence of Adverse events (AEs)
Number of Participants With abnormal Ophthalmic examination | From Day1 to up to Day14
  Change from baseline of ophthalmic examination

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | From Day1 to up to Day14
  Cmax was the highest concentration observed directly from data
Area under the concentration-time curve | From Day1 to up to Day14
  Reflects the actual body exposure to drug after administration of sinlge and multiple dose
Time to Cmax (Tmax) | From Day1 to up to Day14
  Tmax was the time to reach maximum observed plasma concentration
Elimination half-life (t1/2) | From Day1 to up to Day14
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

IPD SHARING:
Plan to Share IPD: No